CLINICAL TRIAL: NCT03276078
Title: A Phase IIa, Open-Label, Repeat-Dose Clinical Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of Aclidinium Bromide/Formoterol Fumarate Fixed Dose Combination Administered Twice-Daily by Inhalation in Chinese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Pharmacokinetics, Safety and Tolerability of Twice-Daily Aclidinium Bromide/Formoterol Fumarate Fixed Dose Combination in Chinese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6572C00001; M-AS464-01 (Other: Clinical Trial Protocol Code)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aclidinium Bromide/Formoterol Fumarate 400/12μg BID (Experimental): Aclidinium bromide/Formoterol Fumarate 400/12μg inhalation powder twice-daily. Oral inhalation via Genuair® dry powder inhaler (DPI).
  Interventions: Drug: Aclidinium Bromide/Formoterol Fumarate 400/12μg BID

INTERVENTIONS:
Drug: Aclidinium Bromide/Formoterol Fumarate 400/12μg BID — Aclidinium bromide/formoterol fumarate 400/12μg administered by inhalation via the Genuair® multidose dry powder inhaler, twice daily (morning and evening) for 5 days

SUMMARY:
A Phase IIa, open-label, repeat-dose trial to investigate the pharmacokinetics (PK), safety and tolerability of single and multiple twice daily doses of inhaled Aclidinium Bromide/Formoterol Fumarate 400/12 μg in 20 Chinese male and female patients with stable moderate to severe COPD.

DETAILED DESCRIPTION:
Screening will be performed within 21 days of dosing on Day 1 at visit 2. Eligible participants will be admitted to the trial center the day preceding the first dosing (day -1).

Participants will receive Aclidinium Bromide/Formoterol Fumarate 400/12 μg twice-daily (morning and evening) on Days 1 to 4. On Day 5 patients will receive the morning dose only. PK and safety assessments will be conducted at specific timepoints on Day 1 to Day 7.

Participants will be discharged 48 h after the last administration of investigational product and completion of the 48-h PK sample collection and safety assessments on Day 7.

A follow-up visit will be performed within 5 days of the last PK sample collection on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate with medical team and staff, willing to participate in the trial, willing to give written informed consent, and comply with the trial procedures and restrictions.
* Chinese men or non-pregnant, non-lactating women, aged ≥40 years old at Visit 1 (Screening).
* Patients with a diagnosis of COPD (GOLD guidelines) for a period of at least 6 months prior to Visit 1 (screening).
* Current or former smokers with a smoking history of ≥10 pack-years.
* Patients with moderate to severe stable COPD (Stage II or Stage III, according to GOLD Guidelines) at Visit 1: post-bronchodilator FEV1 ≥30% and <80% and post-bronchodilator FEV1/FVC <70%.
* Must be able to perform repeatable pulmonary function testing for FEV1 according to ATS/ERS 2005 criteria at Visit 1 (Screening).

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or site staff) or patients employed by or relatives of the employees of the site or sponsor.
* Previous enrolment or randomisation in the present study.
* History or current diagnosis of asthma.
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation (including the mild COPD exacerbation) within 6 weeks prior to screening or during the run-in period.
* Patients hospitalized for COPD exacerbation (an emergency room visit for longer than 24 hours will be considered a hospitalization) within 3 months prior to screening and during the run-in period.
* Use of long-term oxygen therapy ≥15 hours per day.
* Patient with a history of hypersensitivity reaction to inhaled anticholinergics, sympathomimetic amines, inhaled medication, or any component thereof.
* Patients with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention, or patients with symptomatic nonstable prostatic hypertrophy.
* Patients with Type I or uncontrolled Type II diabetes, uncontrolled hypothyroidism or hyperthyroidism, hypokalaemia, hyperadrenergic state, or uncontrolled or untreated hypertension.
* Clinically significant cardiovascular conditions.
* Patient with resting systolic blood pressure ≥160 mmHg, a resting diastolic blood pressure ≥100 mmHg, or a resting heart rate ≤50 bpm or ≥100 bpm at Visit 1 (Screening) or/and at Visit 2 (Day -1 to Day 7).
* Have a body mass index (BMI) ≥40 kg/m2
* Electrocardiogram (ECG) at Screening or Day -1 showing corrected QT interval (QTc) using Fridericia's correction (QTcF) >470 msec.
* Patients with clinically relevant abnormalities in the results of the laboratory tests, ECG parameters (other than QTcF), or in the physical examination at Visit 1, except those related to COPD.
* Positive results for drugs of abuse in the urine at Visit 1 (Screening).
* Positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody and/or human immunodeficiency virus (HIV) I antibodies at Visit 1 (Screening).
* History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer.
* Any other serious or uncontrolled physical or mental condition/disease.
* Patient with a history (within 2 years prior to Visit 1 [Screening]) of drug and/or alcohol abuse that may prevent trial compliance based on investigator judgment.
* Taken any medication within 14 days before the first dose of IP, or hormonal drug products and traditional Chinese medicines within 30 days before the first dose of IP, with the exception of allowed medications listed in the study protocol.
* Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma drawn within 60 days of Day 1 at Visit 2.
* Have participated in a blood/plasma donation or blood loss greater than 400 mL within 90 days or greater than 200 mL within 30 days prior to Visit 1 (Screening).
* Have any clinical condition that might affect the absorption, distribution, biotransformation, or excretion of Aclidinium Bromide/Formoterol Fumarate.
* Have consumed caffeine or any grapefruit-containing products within 48 hours or alcohol within 72 hours before Day -1 at Visit 2.
* Inability to be venipunctured or tolerate venous access as determined by the investigator or designee.
* Inability to use a multidose DPI.
* Subjects unable to give their consent, or subjects of consenting age but under guardianship, or vulnerable subjects.
* In the opinion of the PI, subjects who are unlikely to comply with the protocol requirements, instructions, and trial-related restrictions.
* Previously taken Aclidinium or previously participated in an investigational study of Aclidinium within 6 months of Day 1

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxiang Yu, Principal Investigator — Pneumology Department, The First Hospital of Jilin University
Locations (1):
- Research Site, Changchun, China

REFERENCES:
- [Derived] Zhang H, Daoud SZ, Gillen MS, Calderon N, Heijer M, Molins E, Garcia-Gil E, Chen H, Li Q, Liu C, Ding Y. An Evaluation of the Pharmacokinetics, Safety, and Tolerability of Aclidinium/Formoterol Fixed-Dose Combination Administered in Chinese Patients with Moderate-to-Severe Chronic Obstructive Pulmonary Disease. Drugs R D. 2022 Mar;22(1):35-42. doi: 10.1007/s40268-021-00374-z. Epub 2022 Feb 8. PMID 35133636
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4100&filename=d6572c00001-sap-ed-2_Redacted.pdf
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4100&filename=d6572c00001-pk-csp-v1_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single centre in China. The first participant was enrolled in December 2017 and the last participant visit was in June 2018.
Pre-assignment Details: A total of 97 participants were screened. Of these, 20 were enrolled and received treatment.
Groups:
- AB/FF 400/12 BID: Aclidinium bromide/Formoterol Fumarate 400/12μg inhalation powder twice-daily. Oral inhalation via Genuair® dry powder inhaler (DPI).
Period: Overall Study
Arm/Group | AB/FF 400/12 BID
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Includes all participants who received at least one dose of investigational product.
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Single Dose).
Description: Observed maximum concentration, taken directly from the individual concentration-time curve (first dose).
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post the morning dose on Day 1
Population: Pharmacokinetic analysis set: All participants who took at least one dose of the IP and had at least one of the parameters (Cmax, Css,max, AUC, AUClast or AUCss,tau) evaluable and were assumed not to be affected by factors such as important protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
pg/mL
  Aclidinium Bromide | 45.82 (84.54)
  LAS34850 | 3149 (55.56)
  LAS34823 | 38.82 (86.60)
  Formoterol Fumarate | 4.786 (62.78)

2. Primary Outcome: Tmax of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Single Dose).
Description: Time to maximum concentration (h), taken directly from the individual concentration-time curve (first dose).
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post the morning dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
hours
  Aclidinium Bromide | 0.08 [0.08 to 0.50]
  LAS34850 | 3.00 [1.50 to 6.00]
  LAS34823 | 1.75 [0.08 to 4.00]
  Formoterol Fumarate | 1.00 [0.08 to 3.00]

3. Primary Outcome: Cmin of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Single Dose).
Description: Minimum plasma drug concentration at the end of the dosing interval (first dose), where possible.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post the morning dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
pg/mL
  Aclidinium Bromide Not calculable | 0 (0)
  LAS34850 | 627.7 (52.02)
  LAS34823 Not calculable | 0 (0)
  Formoterol Fumarate Not calculable | 0 (0)

4. Primary Outcome: AUC(Last) of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Single Dose).
Description: Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post the morning dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hour/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
pg*hour/mL
  Aclidinium Bromide | 78.61 (90.69)
  LAS34850 | 20280 (54.28)
  LAS34823 | 201.1 (106.3)
  Formoterol Fumarate | 20.04 (64.22)

5. Primary Outcome: AUC(Tau) of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Single Dose).
Description: Area under the plasma concentration curve during the first dosing interval, tau (first dose).
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post the morning dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hour/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
pg*hour/mL
  Aclidinium Bromide | 85.45 (79.02)
  LAS34850 | 20330 (54.24)
  LAS34823: number analyzed (Participants) | 18
  LAS34823 | 252.9 (60.63)
  Formoterol Fumarate: number analyzed (Participants) | 19
  Formoterol Fumarate | 22.78 (43.64)

6. Primary Outcome: Css,Max of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Observed maximum concentration, taken directly from the individual concentration-time curve at steady state.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
pg/mL
  Aclidinium Bromide | 60.86 (150.0)
  LAS34850 | 3691 (56.03)
  LAS34823 | 81.02 (69.52)
  Formoterol Fumarate | 6.465 (84.34)

7. Primary Outcome: Css,Min of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Observed minimum concentration, taken directly from the individual concentration-time curve within a dosing interval on Day 5.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
pg/mL
  Aclidinium Bromide | 4.528 (47.34)
  LAS34850 | 1032 (43.05)
  LAS34823 | 22.88 (47.22)
  Formoterol Fumarate | 1.281 (36.63)

8. Primary Outcome: Tss,Max of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Time to maximum concentration (h), taken directly from the individual concentration-time curve at steady state.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
hours
  Aclidinium Bromide | 0.08 [0.08 to 0.50]
  LAS34850 | 3.00 [0.08 to 4.00]
  LAS34823 | 0.50 [0.08 to 3.00]
  Formoterol Fumarate | 0.08 [0.08 to 1.50]

9. Primary Outcome: λz of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Terminal rate constant, estimated by log-linear least square regression of the terminal part of the concentration-time curve.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
1/hours
  Aclidinium Bromide | 0.053 (0.040)
  LAS34850 | 0.045 (0.018)
  LAS34823 | 0.048 (0.021)
  Formoterol Fumarate | 0.057 (0.029)

10. Primary Outcome: t½λz of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Terminal half-life (h), estimated as (ln2)/λz.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
hours
  Aclidinium Bromide | 19.42 (11.10)
  LAS34850 | 20.95 (18.78)
  LAS34823 | 17.34 (8.096)
  Formoterol Fumarate | 14.06 (4.796)

11. Primary Outcome: AUC(ss,Tau) of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Area under the plasma concentration curve during the dosing interval, tau at steady state.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hour/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
pg*hour/mL
  Aclidinium Bromide | 168.8 (82.15)
  LAS34850 | 27300 (52.29)
  LAS34823 | 540.9 (54.97)
  Formoterol Fumarate | 31.98 (51.60)

12. Primary Outcome: CL/F of Aclidinium Bromide and Formoterol Fumarate (Multiple Doses).
Description: Apparent plasma clearance for parent drug estimated as dose divided by AUCss
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
L/hour
  Aclidinium Bromide | 3140 (2868)
  Formoterol Fumarate | 422.2 (222.7)

13. Primary Outcome: Vz/F of Aclidinium Bromide and Formoterol Fumarate (Multiple Doses).
Description: Apparent volume of distribution for parent drug at terminal phase, estimated by dividing the apparent clearance (CL/F) by λz.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
L
  Aclidinium Bromide | 81990 (87200)
  Formoterol Fumarate | 8284 (5161)

14. Primary Outcome: Cav of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Average plasma concentration during a dosing interval, estimated as AUC(ss,tau)/12
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
pg/mL
  Aclidinium Bromide | 14.07 (82.15)
  LAS34850 | 2275 (52.29)
  LAS34823 | 45.07 (54.97)
  Formoterol Fumarate | 2.665 (51.60)

15. Primary Outcome: %Fluctuation of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Fluctuation index during a dosing interval estimated as 100*(Cmax-Cmin)/Cav (%).
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
Percentage
  Aclidinium Bromide | 452.5 (269.4)
  LAS34850 | 117.0 (24.69)
  LAS34823 | 132.0 (57.81)
  Formoterol Fumarate | 205.9 (90.94)

16. Primary Outcome: Rac(Cmax) of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Accumulation ratio for Cmax estimated as Css,max on Day 5/Cmax on Day 1
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
ratio
  Aclidinium Bromide | 1.297 (216.6)
  LAS34850 | 1.185 (80.29)
  LAS34823 | 2.070 (113.5)
  Formoterol Fumarate | 1.384 (90.21)

17. Primary Outcome: Rac[AUC(Tau)] of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Accumulation ratio for AUC(tau) estimated as AUC(ss,tau) on Day 5/AUC(tau) on Day 1
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
ratio
  Aclidinium Bromide | 1.966 (108.9)
  LAS34850 | 1.355 (76.54)
  LAS34823: number analyzed (Participants) | 17
  LAS34823 | 2.157 (82.00)
  Formoterol Fumarate: number analyzed (Participants) | 18
  Formoterol Fumarate | 1.436 (56.27)

18. Primary Outcome: Rac(Cmin) of Aclidinium Bromide, Its Metabolites and Formoterol Fumarate (Multiple Doses).
Description: Accumulation ratio for Cmin estimated as Css,min on Day 5/Cmin on Day 1.
  Additional parameters may be determined where appropriate.
Time Frame: Pre-dose and 5, 15, and 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post the morning dose on Day 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 19
ratio
  Aclidinium Bromide: number analyzed (Participants) | 3
  Aclidinium Bromide | 1.877 (45.19)
  LAS34850 | 1.641 (69.91)
  LAS34823: number analyzed (Participants) | 14
  LAS34823 | 2.601 (54.86)
  Formoterol Fumarate: number analyzed (Participants) | 12
  Formoterol Fumarate | 1.822 (31.43)

19. Secondary Outcome: Adverse Events (AEs)/Serious AEs (SAEs)
Description: Assessment of the safety in terms of the incidences of AEs/SAEs after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants
  Any AE | 5
  Any SAE | 1

20. Secondary Outcome: Treatment-emergent AEs Related to Blood Pressure
Description: Assessment of the safety in terms of notable changes from baseline in blood pressure after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants
  Blood pressure increased | 1

21. Secondary Outcome: Treatment-emergent AEs Related to Clinical Laboratory Parameters (Haematology)
Description: Assessment of the safety in terms of haematology parameters after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants | 0

22. Secondary Outcome: Treatment-emergent AEs Related to Clinical Laboratory Parameters (Urinalysis)
Description: Assessment of the safety in terms of urinalysis parameters after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants
  Urine protein present | 3
  Haematuria | 1

23. Secondary Outcome: Treatment-emergent AEs Related to Clinical Laboratory Parameters (Serum Biochemistry)
Description: Assessment of the safety in terms of serum biochemistry parameters (Alanine aminotransferase [ALT], Aspartate aminotransferase [AST], alkaline phosphatase [ALP], Gamma-glutamyl transferase [GGT], bilirubin, creatine kinase, lactate dehydrogenase, urea nitrogen, creatinine, urate, cholesterol, glucose, sodium, potassium, calcium, chloride, phosphate, protein, and albumin) after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants | 0

24. Secondary Outcome: Treatment-emergent AEs Related to 12-lead ECG Parameters
Description: Assessment of the safety in terms of the 12-lead ECG parameters after administration of Aclidinium Bromide/Formoterol Fumarate 400/12 μg BID for 5 days.
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Population: Safety analysis set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AB/FF 400/12 BID
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Screening (Day -21) to Follow-up visit (Days 8-12)
Description: The Safety population included all participants who received at least one dose of investigational product.
  AE summary includes treatment-emergent AEs, that is AEs starting after the first administration of investigational product, until 15 days from last dose.
Arm/Group | AB/FF 400/12 BID
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 BID (N=20)
Bronchitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 BID (N=20)
Protein urine present (Investigations) | 3 (3)

LIMITATIONS AND CAVEATS:
A possible limitation of the study is the high between-participant variability, which was likely related to suboptimal inhalation technique in many participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and / or presentation whether complete or partial, of any part of the data or results of this study will not be allowed until global publication and study results disclosure by the sponsor as per EMA / FDA regulatory compliance obligations, and only after mutual agreement between the Investigator and AstraZeneca

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03276078/SAP_000.pdf
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03276078/Prot_001.pdf